CLINICAL TRIAL: NCT03364699
Title: High-EPA and High-DHA Fish Oils and Soybean Lecithin Modulate Inflammation and Neutrophil Properties in Runners Before and After a Half-marathon
Brief Title: Fish Oils and Soybean Lecithin Supplementation Modulate Immune Function in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Tania Cristina Pithon-Curi, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 979/2010
Record Dates: First submitted 2017-01-03; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Immune Dysfunction
Keywords: strenuous exercise; dietary supplementation; immune system; leucocyte function; inflammation
MeSH Terms: conditions — Immune System Diseases; Inflammation | interventions — Dietary Supplements; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dietary supplementation (Active Comparator): The volunteers ingested 3 g daily of Soybean lecithin or fish oil rich in docosa-hexanoic acid (DHA) containing 1.5 g DHA and 0.3 g EPA (DHA:EPA = 5:1) or fish oil rich in eicosapentaenoic acid (EPA) containing 1.6 g EPA and 0.3 g DHA (EPA:DHA = 5.4:1) during 60 days.
  Interventions: Dietary Supplement: dietary supplementation
- Exercise (Experimental): All volunteers performed two half-marathons. In the first half-marathon, all participants were not supplemented. In the second half-marathon, participants were supplemented. Blood samples were collected before and after both half-marathon race.
  Interventions: Dietary Supplement: dietary supplementation; Other: Exercise

INTERVENTIONS:
Dietary Supplement: dietary supplementation — The volunteers ingested 3 g daily of Soybean lecithin or fish oil rich in docosa-hexanoic acid (DHA) containing 1.5 g DHA and 0.3 g EPA (DHA:EPA = 5:1) or fish oil rich in eicosapentaenoic acid (EPA) containing 1.6 g EPA and 0.3 g DHA (EPA:DHA = 5.4:1) during 60 days.
Other: Exercise — All volunteers performed two half-marathons. In the first half-marathon, all participants were not supplemented. In the second half-marathon, all participants were supplemented. Blood samples were collected before and after both half-marathon race.
  Arms: Exercise

SUMMARY:
The purpose of this study was evaluate the comparative effects of FO rich in EPA (FO-EPA) and FO rich in DHA (FO-DHA) on inflammation and neutrophil properties after a prolonged and strenuous exercise. The effect of soybean lecithin on the same parameters and conditions also was evaluated.

DETAILED DESCRIPTION:
The volunteers were not taking any medication during the study. All individuals signed an informed consent form to the study protocol. Both experimental procedure and informed consent form of this study were in accordance with Guide for the Care and Use of Humans.

All volunteers performed two half-marathons. In the first half-marathon, all participants were not supplemented. Dietary supplementation was initiated immediately after the first race. The volunteers were randomly separated into 3 groups: Soybean lecithin group; Fish oil-DHA group and Fish oil-EPA group. The volunteers ingested 3 g daily of SL or FO-DHA containing 1.5 g DHA and 0.3 g EPA or FO-EPA containing 1.6 g EPA and 0.3 g DHA (EPA:DHA = 5.4:1) during 60 days.

Experimental design:

First race - not supplemented, blood samples were collected before (Phase I) and immediately after race (Phase II).

Second race - dietary supplemented, blood samples were collected before (Phase III) and immediately after the race (Phase IV).

Results were analyzed by two-way analysis of variance (two-way ANOVA) and Tukey post-hoc test. The statistical analysis of the half-marathon effect was performed using nonparametric t tests. Results were considered statistically significant for P<0.05.

ELIGIBILITY:
Inclusion Criteria:

Healthy recreational half-marathon runners.

Exclusion Criteria:

Auto-immune disease Inflammatory disease Cardiorespiratory disease

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Neutrophil expression of ICAM-1, L-selectin, FasR and TRAIL | Immediately after the first race (Phase II) and immediately after the second race in supplemented athletes (Phase IV).
  Neutrophil expression was expressed in fluorescence intensity evaluated by flow cytometry at 530/30 nm (FITC) 660/20 nm (APC) or 695/40 nm (PE) wavelengths (BD Accuri cytometer).

SECONDARY OUTCOMES:
Plasma concentrations of IL-1beta, IL-4, IL-6, IL-8, IL-10, and TNF-alpha. | Immediately after the first race (Phase II) and immediately after the second race in supplemented athletes (Phase IV).
  Plasma concentrations of IL-1beta, IL-4, IL-6, IL-8, IL-10, and TNF-alpha in pg/mL were measured by Millipore® Multiplex Assays Using Luminex® (Millipore Corp., MA).

OTHER OUTCOMES:
Blood leukocytes counts | Immediately after the first race (Phase II) and immediately after the second race in supplemented athletes (Phase IV).
  Blood leukocyte counts in number of cells per mL was performed immediately after collection using routine automated system (hematological analysis cytochemic/isovolumetric assay).
Plasma LDH activity | Immediately after the first race (Phase II) and immediately after the second race in supplemented athletes (Phase IV).
  Plasma lactate dehydrogenase (LDH) activity in U/L was immediately measured using an automated system (kinetic-enzymatic assay).

CONTACTS AND LOCATIONS:
Overall Officials: Tania C Pithon-Curi, PhD, Principal Investigator — University of Sao Paulo and Cruzeiro do Sul University
Locations (1):
- Cruzeiro do Sul University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No